CLINICAL TRIAL: NCT04910737
Title: Safety and Effectiveness of Extended Circumferential Decompression for Thoracic Ossification of Posterior Longitudinal Ligament：a Single-center Experience
Brief Title: Safety and Effectiveness of Extended Circumferential Decompression for Thoracic Ossification of Posterior Longitudinal Ligament
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-439
Record Dates: First submitted 2021-05-28; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Indications and Effectiveness for Extended Posterior Circumferential Decompression
Keywords: circumferential decompression; thoracic ossification of posterior longitudinal ligament; kyphosis; neurological outcomes
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: extended posterior circumferential decompressive surgery — After the pedicle screws were implanted, laminectomy was performed. Kyphotic correction was done through a temporary rod to reduce the tension of spinal cord. The posterior 1/3 of the vertebral body was resected using a high-speed drill, preserving the anterior wall of the spinal canal to protect the cord from disturbance. The dissection of adhesion at the anterior side of spinal cord was to be done through a posterolateral direction. The region of posterior resection was expanded, including bilateral residual articular processes, transverse processes and pedicles. Slightly press down the ossified lesion, and detach it from the dura mater (perform a sharp dissection if necessary) followed by completely removal. If cerebrospinal fluid leakage was encountered during the process, autologous fat, fascia or gelatin sponge can be applied locally for packaging.

SUMMARY:
The study was to evaluate the indications, efficiency and safety of the extended posterior circumferential decompression technique for the treatment of thoracic ossification of posterior longitudinal ligament (TOPLL) with dura adhesions or ossification.

DETAILED DESCRIPTION:
The clinical characteristics of patients with TOPLL combined with dura adhesions who underwent extended circumferential decompression in our hospital were retrospectively investigated. TOPLL adhered with dura matter or dura ossification were detected intraoperatively in all the cases. Imaging evaluation included the ossification-kyphosis angle and the fixed-segment kyphosis angle. A modified Japanese Orthopedic Association Score (JOA score) was applied for the evaluation of clinical outcomes.

ELIGIBILITY:
Inclusion Criteria: (1) thoracic myelopathy caused by TOPLL with or without TOLF; (2) severe adhesions between dura mater and ossified lesion with or without dura ossification confirmed intraoperatively; (3) extended posterior circumferential decompression was applied; (4) pedicle screw instrumentations were implanted after decompression; (5) follow-up for more than 6 months; (7) complete clinical data.

Exclusion Criteria:

(1) spinal deformities; (2) thoracic spine fractures; (3) syringomyelia, spinal tumor, myelitis, etc.; (4) coexisted with cervical spondylosis and lumbar stenosis; (5) post operation of thoracic spinal stenosis; (6) recurrent myelopathy caused by lesions in other levels than the decompressed segments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No limit
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
A modified Japanese Orthopedic Association Score | 2 years
  Spinal neurological function evaluation by Japanese Orthopedic Association

CONTACTS AND LOCATIONS:
Overall Officials: Ruofu Tang, Study Director — Second affiliated hospital of medicine, Zhejiang University
Locations (1):
- Second affiliated hospital of Zhejiang University, School of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No